CLINICAL TRIAL: NCT03980847
Title: Teh Histomorphometric Study of Nanocrystalline Hydroxyapatite (Nano Bone) Wif Alendronate in Teh Preservation of Teh Tooth Socket
Brief Title: Evaluation, the Histomorphometric Study of Nanocrystalline Hydroxyapatite (Nano Bone) Wif Alendronate in the Preservation of the Tooth Socket
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Islamic Azad University, Sanandaj (Other)
Responsible Party: Principal Investigator, Amirhossein Farahmand, assistant prof, Islamic Azad University, Sanandaj
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2036
Record Dates: First submitted 2019-05-13; First posted 2019-06-10 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Bone Resorption
MeSH Terms: conditions — Bone Resorption | interventions — Alendronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alendronate 20 mg with bone graft (Active Comparator): after tooth extraction, put teh Alendronate 20mg with bone graft within teh tooth socket
  Interventions: Drug: Alendronate 20 mg
- bone graft alone (Active Comparator): after tooth extraction, put the bone graft within the tooth socket
  Interventions: Drug: Alendronate 20 mg; Procedure: Nanocrystal hydroxyapatite

INTERVENTIONS:
Drug: Alendronate 20 mg — The Alendronate 20 mg combined with nanocrystalline hydroxyapatite as a synthetic bone substitute for socket preservation after tooth extraction
  Other Names: Group A
Procedure: Nanocrystal hydroxyapatite — Postextraction Sockets Preserved With Nanocrystal hydroxyapatite as a synthetic bone substitute alone as a bone graft
  Other Names: Group B
  Arms: bone graft alone

SUMMARY:
Twenty patients referring to periodontics department of Boroujerd Azad university of dentistry after obtaining consent to participate in teh research project, which TEMPhas more TEMPthan 20 teeth, are over 18 years old and require socket preservation surgery to tooth extraction for teh periodontal problem, caries or Fractures were selected.

DETAILED DESCRIPTION:
20 healthy patients referring to periodontics department of Boroujerd Azad university of dentistry after obtaining consent to participate in the research project, which has more than 20 teeth, are over 18 years old and require socket preservation surgery to tooth extraction for the periodontal problem, caries or Fractures were selected. Furthermore, divided the socket randomly to two groups(A, B)including A: bone graft wif Alendronate and B: bone graft alone, after 3 months wif trephine will collect the samples. following the histomorphometric analysis.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years old
2. tooth fracture, root caries
3. Patients are volunteered for placement of teh implant

Exclusion Criteria:

1. systemic diseases
2. Pregnancy and breastfeeding
3. malignancy, radiation therapy,
4. history of periodontal surgery during teh six months ago.
5. medicine(phosphonates, antibiotic,...)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
New bone formation (bone area as percent) | 3 month
  Combination Lovastatin produced increased vital bone more percentage compared to the nanocrystal bone graft alone group. The new bone formation and alveolar ridge preservation with bone graft after extraction of pre-molar teeth could result in the maintenance of sufficient bone volume to place an implant in an ideal restorative position without the need for auxiliary implant site development procedures.

CONTACTS AND LOCATIONS:
Locations (1):
- Amirhossein Farahmand, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No